CLINICAL TRIAL: NCT00444561
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Multicenter Exploratory Study to Evaluate Various Pharmacodynamic Effects of Subcutaneously Infused or Injected Pramlintide in Obese Subjects
Brief Title: Exploratory Study to Evaluate Various Pharmacodynamic Effects of Subcutaneously Infused or Injected Pramlintide in Obese Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 137-160
Record Dates: First submitted 2007-03-06; First posted 2007-03-08 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-05

CONDITIONS: Overweight; Obesity
Keywords: pramlintide; Symlin; Amylin
MeSH Terms: conditions — Overweight; Obesity | interventions — pramlintide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pramlintide acetate (AC137) (Active Comparator): Pramlintide acetate (AC137) injection is a clear, colorless, sterile solution for SC administration. It consists of pramlintide in sodium acetate buffer, pH 4.0, containing 43 mg/mL mannitol as an osmolality modifier and 2.25 mg/mL metacresol as a preservative. The concentration of pramlintide injection to be used in this study is 0.6 mg/mL.
  Interventions: Drug: pramlintide acetate

INTERVENTIONS:
Drug: pramlintide acetate — Clear, colorless, sterile solution for SC administration

SUMMARY:
This exploratory study is designed to evaluate various pharmacodynamic effects of subcutaneously (SC) infused or injected pramlintide in obese, nondiabetic male and postmenopausal female (not on hormone replacement therapy) subjects. The study will also assess the safety and tolerability of pramlintide administered by SC infusion or injection.

ELIGIBILITY:
Inclusion Criteria:

* Is <6'3" (190.5 cm) tall and weighs <300 lb (~136.3 kg)
* Is obese with a body mass index (BMI) >=30 kg/m^2 to <=45 kg/m^2 and with a history consistent with progressive weight gain and development of obesity not secondary to drastic or traumatic initiating events (e.g., excessive weight gain due to cessation of smoking)
* Is a nonsmoker (never smoked or has not smoked for at least 2 years)
* Does not have a clinical diagnosis of diabetes
* Has not had a major change in daily physical activity within 2 months prior to study start (e.g., initiation of an exercise program)
* Usually consumes three major meals (morning, midday, and evening) each day and rarely (less than once a week) wakes up to eat during the night

Exclusion Criteria:

* Is currently enrolled in a weight loss program or plans to enroll in a weight loss or exercise program within the next 3 months
* Is currently treated or expected to require or undergo treatment or has been treated within 2 months before screening with medications that are excluded:

  * Over the counter antiobesity agents including herbal supplements or prescription antiobesity agents approved for the long-term (including orlistat [Xenical] and sibutramine [Meridia]) and the short-term (including phentermine [Adipex-P, Celltech, Pro-Fast SA, Pro-Fast SR, Fastin, Oby trim, Zantryl, Teramine, Phentride, Phentercot, Obephen, Oby-cap], mazindol [Sanorex and Mazanor], methamphetamine [Desoxyn], diethylpropion [Tenuate and Tenuate Dospan], phendimetrazine [Bontril, Prelu-2, Melfiat 105, Unicelles, X-Trozine, Plegine, Adipost, Obezine, Phendiet-105, PT 105] and benzphetamine [Didrex]) treatment of obesity
  * Systemic steroids by oral, intravenous, or intramuscular route or potent topical steroids that are known to result in high systemic absorption
  * Alpha- or Beta-Blockers, centrally acting sympathicolytic or sympathicomimetic agents, reserpin, guanethidine, etc.
  * Psychotropic medications (e.g., tricyclic antidepressants, monoamine oxidase [MAO] inhibitors, selective serotonin reuptake inhibitors [SSRIs], neuroleptics, lithium, and benzodiazepines)
  * Hypnotic-sedative medications or medications that may affect sleeping behavior including medications containing caffeine
  * Drugs that directly affect gastrointestinal motility, including but not limited to: metoclopramide (Reglan®) and cisapride (Propulsid®); and macrolide antibiotics such as erythromycin and newer derivatives
* Has received any investigational drug within 3 months before study start
* Has participated previously in a study using pramlintide

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 184 (Actual)
Dates: Start 2004-08; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
To evaluate various pharmacodynamic effects (including effects on body weight, food intake, and other parameters) of subcutaneously (SC) infused or injected pramlintide in obese subjects. | 73 Days

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of SC infused or injected pramlintide in obese subjects. | 73 Days

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Porter, MD, Study Director — Amylin Pharmaceuticals, LLC.
Locations (10):
- United States (10):
  - Research Site, Chula Vista, California
  - Research Site, Long Beach, California
  - Research Site, San Diego, California
  - Research Site, DeLand, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Lexington, Kentucky
  - Research Site, Baton Rouge, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Butte, Montana
  - Research Site, San Antonio, Texas